CLINICAL TRIAL: NCT04935242
Title: Evaluation of the Modalities of Administration of Synthetic Oxytocin During Spontaneous Labor
Acronym: LAMA
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: LAMA (LAbour Management)
Record Dates: First submitted 2021-06-15; First posted 2021-06-22 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Oxytocin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Syntocinon was granted marketing authorization in France in 1970. Since the 1960s, it has been frequently used during childbirth, particularly in cases of stagnation of cervical dilatation due to a lack of uterine contractility. According to the latest National Perinatal Survey of 2010, 66.5% of patients go into labor spontaneously and 58% of them receive Syntocinon during labor.

The reported maternal effects associated with the use of synthetic oxytocin include uterine hyperactivity, postpartum hemorrhage (PPH) and severe PPH. The administration of oxytocin increases the risk of uterine hyperactivity in a dose-dependent manner. Regarding fetal risk, the reported adverse effects concern fetal heart rate abnormalities related to uterine hyperactivity. However, no study has shown an association between oxytocin administration and excess neonatal morbidity and mortality, except in the subpopulation of patients with a scarred uterus.

DETAILED DESCRIPTION:
In the 1950s, the speed of cervical dilation during labor was studied by Friedman. Dilatation is then divided into several phases:

* A first phase known as the latency phase which corresponds to the effacement of the cervix and its dilation up to 3 cm. It lasts on average 7 hours for a primipara and 5 hours for a multipara.
* A second active phase which corresponds to the dilation of the effaced cervix. This phase includes the progressive acceleration phase (up to 4-5 cm of dilation), a phase of maximum slope (up to 9 cm) and a deceleration phase where the slope decreases from 9 cm to full dilation (FD). This active phase lasts, on average, 4h30 in primiparous women and 2h30 in multiparous women.

Friedman concluded that cervical dilatation should be of the order of 1.5 cm/h and more in the active phase and that it should not fall below 1 cm/h in nulliparous women and 1.5 cm/h in multiparous women.

In the 1980s, the use of syntocinon became commonplace.Under the influence of an Irish physician, O'Driscoll, policies of quasi-systematic direction of labor were implemented, in particular in nulliparous women. This concept of active management of labor was developed in response to the observation of a high rate of cesarean sections performed for stagnation. This active labor management included systematic rupture of membranes (amniotomy) and infusion of Syntocinon when the dilation rate was less than 1 cm/h.

Beginning in the 2000s, Zhang also focused on the physiological duration of labor. He showed that a so-called normal labor could be much longer than previously described, especially before 6cm of cervical dilation. In 2010, he proposed a new partogram for nulliparous patients.

Finally, Neal performed a review of the literature in 2010, evaluating 7,009 low risk primiparous patients in spontaneous labor. He showed longer active phase durations than those described so far. The duration of labor at the 95th percentile was 13.4 hours and the average dilation rate around 0.6cm/h. The author concludes that a dilation speed of 0.5 cm/h can be tolerated in primiparous patients, without requiring additional intervention.

In this context, new French recommendations regarding oxytocin administration during spontaneous labor were published in December 2016. These recommendations were based mainly on studies including patients at term, without a history of cesarean section, with a single-fetal pregnancy and cephalic presentation:

* It is recommended that the diagnosis of abnormal progression of labor (dynamic dystocia) not be made before 5-6 cm of cervical dilation, corresponding to the end of the latency phase of the 1st stage of labor (professional agreement).
* It is recommended to consider a dilation speed as abnormal if it is less than 1 cm/4 h between 5 and 7 cm, and less than 1 cm/2 h beyond 7 cm of dilation (grade B)
* In the absence of dynamic dystocia, active direction of labor is not recommended (Grade B)
* Before 5 cm, it is recommended that neither amniotomy nor oxytocin administration be performed routinely, regardless of the speed of dilation (Grade B)
* Early epidural analgesia (EAP) during the latent phase does not increase the frequency of indications for oxytocin administration during spontaneous labor (Grade B).
* If dynamic dystocia is present during the active phase, amniotomy is recommended before oxytocin administration (professional agreement).
* If the 2nd stage is prolonged beyond 2 hours, it is recommended that oxytocin be administered to correct a lack of progression of presentation (professional agreement)
* It is recommended to start at an initial dose of 2 mIU/min (professional agreement).
* Intervals of at least 30 min are recommended before each oxytocin dose increase (Grade B).
* It is recommended that oxytocin be increased in dose increments of 2 mIU/min, not to exceed an absolute rate of 20 mIU/min, and that dose escalation be discontinued when cervical change or 5 uterine contractions per 10 min are achieved (professional consensus).

These recommendations began to be applied in the maternity ward of Saint Joseph Hospital following their publication, starting in January 2017. These recommendations concern patients at low obstetrical risk, i.e., presenting a singleton pregnancy with a fetus estimated to be eutrophic and in cephalic presentation, a non-scarring uterus and spontaneous labor at term.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Single pregnancy
* Non-scarring uterus
* Fetus estimated to be eutrophic in prenatal
* Cephalic presentation
* Spontaneous labor from 37 weeks of amenorrhea

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient objecting to the use of her data for this research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who delivered at Paris Saint Joseph Hospital in 2016 and 2018
Sampling Method: Non-Probability Sample
Enrollment: 3311 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2021-09-19 (Actual); Study Completion 2022-04-26 (Actual)

PRIMARY OUTCOMES:
Assessment of professional practices before the recommendations for clinical practice (RPC) published in December 2016, concerning the modalities of administration of synthetic oxytocin during physiological labor | Day 1
  Difference in management modalities between two groups of patients:
  * A first group of patients who gave birth in 2016
  * A second group of patients who gave birth in 2018
Assessment of professional practices after the recommendations for clinical practice (RPC) published in December 2016, concerning the modalities of administration of synthetic oxytocin during physiological labor | Day 1
  Difference in management modalities between two groups of patients:
  * A first group of patients who gave birth in 2016
  * A second group of patients who gave birth in 2018

SECONDARY OUTCOMES:
Evaluation of the impact of the application of the new recommendations on the rate of vaginal deliveries | Day 1
  Difference between these two groups of patients in terms of rate of vaginal delivery
Evaluation of the impact of the application of the new recommendations on the rate of postpartum hemorrhage | Day 1
  Difference between these two groups of patients in terms of rate of postpartum hemorrhage
Evaluation of the impact of the application of the new recommendations on the rate of neonatal morbidity | Day 1
  Difference between these two groups of patients in terms of rate of average APGAR scores in newborns measured at 1, 5 and 10 minutes of life

CONTACTS AND LOCATIONS:
Overall Officials: Johan PACELLI, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France